CLINICAL TRIAL: NCT00953342
Title: Impact of Aerobic Exercise on Asthma Morbidity
Acronym: Ex-Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Simon Bacon, Researcher, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOP93807
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2016-06

CONDITIONS: Asthma
Keywords: AEROBIC EXERCISE; ASTHMA CONTROL; ASTHMA QUALITY OF LIFE; INFLAMMATION; TREATMENT
MeSH Terms: conditions — Asthma; Inflammation | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic exercise (Experimental): 12 weeks of supervised aerobic exercise and standard care
  Interventions: Behavioral: Aerobic exercise
- Usual care (Placebo Comparator): 12 weeks of standard care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Aerobic exercise — 12 weeks of supervised exercise, 3 x week, 1 hour sessions
  Arms: Aerobic exercise
Behavioral: Usual care — Standard medical care
  Arms: Usual care

SUMMARY:
Asthma is a chronic disorder of the airways primarily driven by increased airway inflammation, and is an escalating medical problem in Canada. For example, between 1994 and 2001 there was a 40% increase in the number of Canadians who had asthma. Not only is the prevalence of asthma increasing but there has been a rapid rise in the number of asthma events and costs associated with asthma and poor asthma control. It has been estimated that the global cost of caring for asthma exceeds that of AIDS/HIV and tuberculosis combined. These increases have occurred in spite of the development of clear asthma management guidelines. There is evidence to suggest that aerobic exercise, e.g., running or cycling, may improve asthma symptoms and control in children. However, there are currently no studies that have systematically assessed the effects of exercise on asthma control or symptoms in adults. The current proposed study will assess the effects of aerobic exercise in sedentary patients with poorly controlled asthma. In addition to usual medical care, 52 patients will participate in a supervised aerobic exercise program. The program will consist of 3 X 1hr sessions of supervised exercise per week for 12 weeks. Another 52 patients will only maintain usual medical care. The asthma control, quality of life, and inflammatory profile will be evaluated at baseline and following the 12 weeks of treatment. The investigators believe that: (1) The exercise intervention will significant improve asthma control and asthma quality of life; (2) The exercise intervention will result in significant improvements in inflammatory profiles; and (3) These changes in the inflammatory profile will be directly related to the improvements in asthma control and quality of life.

DETAILED DESCRIPTION:
Introduction: Asthma is a chronic respiratory disorder primarily driven by increased airway inflammation. It is one of the most prevalent chronic conditions affecting Canadians. It is the most common chronic illness affecting children and the fourth most common disorders affecting adults. In 2001, nearly 2.2 million (8.4%) Canadians were diagnosed as having asthma. More importantly, asthma is an escalating medical problem in Canada, e.g., between 1994 and 2001, there was a 40% increase in the number of Canadians with asthma. Not only is the prevalence of asthma increasing, but there has been a rapid rise in the morbidity and costs associated with asthma and its poor control. The WHO estimated that the global cost of caring for asthma exceeds that of AIDS/HIV and tuberculosis combined. Though recent guidelines have emphasized the importance of improving asthma control and quality of life, leading to huge amounts of resource being dedicated to this, more than 50% of adult patients with asthma remain poorly controlled. As current treatment strategies appear to be failing, it is important to target simple, cost effective interventions that are applicable for most patients with asthma and will increase overall levels of control and decrease asthma morbidity. There is evidence to suggest that aerobic exercise may improve asthma symptoms and control in children. In addition, there is evidence that exercise directly improves inflammatory and immune profiles in non-asthma patients, which may provide the mechanism by which exercise could improve asthma. However, there are no known studies that have systematically assessed the effects of aerobic exercise on asthma control, quality of life or immune function in adult asthma populations.

Objective: The primary objective of the current application is to assess the efficacy of aerobic exercise as an intervention to improve asthma control and quality of life in adult patients with asthma. The results of this study will provide data that will inform physicians and members of the Thoracic community about the benefits of exercise for asthma. The study will also assess potential inflammatory pathways by which exercise may elicit improvements in asthma morbidity. The results of this study should be available for the next Canadian Thoracic Society Canadian Adult Consensus Guidelines.

Methodology: The current proposal is for a study of aerobic exercise in sedentary patients with poorly controlled asthma. In addition to usual care, 52 patients will undertake supervised aerobic exercise. The exercise program will consist of 3 X 1hr sessions of supervised exercise per week for 12 weeks. The exercise routine, under medical supervision, will consist of 10 minutes of warm up exercises, 40 minutes of biking and/or walking (and eventually jogging), and 10 minutes of cool down exercises. These patients will be compared to a group of 52 patients who will follow their usual regimen, this group will be offered the exercise programme once they have completed the post assessments. For the primary outcomes (asthma control [Asthma Control Questionnaire], quality of life [Asthma Quality of Life Questionnaire]) and secondary outcomes (inflammatory profile) will be evaluated at baseline and after 12 weeks (the length of the treatment). To check the efficacy of the intervention both lung function, ambulatory peak flow, and exercise tolerance data will also be collected. Repeated measures analysis of covariance-type models with time (pre, post intervention) as the within subject factor, group (exercise, usual care) as the between factor, and sex, age, and asthma severity as the covariates will be used for the primary outcome variables. To assess the potential mechanistic role of inflammation on the exercise-asthma relationship a series of regression-like GLMs will be conducted.

It is hypothesized that: (1) The exercise intervention will result in clinically and statistically significant improvements in levels of asthma control and asthma quality of life; (2) The exercise intervention will result in clinically and statistically significant improvements in inflammatory profiles, with reductions in Th2 cytokines, and activation of inflammatory cells, and increases in Th1 cytokines; and (3) Changes in inflammatory profile will be directly linked to improvements in asthma measures.

We believe that the proposal will have great clinical significance for patient management. This project will be the first to systematically evaluate the benefits of exercise training on asthma control and quality of life in adult asthma patients. We anticipate that the results of this study will form the basis for new national and international guidelines and will provide an evidence-based background for physicians to prescribe aerobic exercise for patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed asthma (confirmed by medical record evidence of bronchodilator reversibility of 12% or a minimum of 180 cc or PC20 methacholine <= 16 mg/ml)
* Sedentary (currently do less than 60 min of structured / planned physical activity per week)
* Taking at least 250 mg fluticasone equivalent per day
* On stable dose and regimen of asthma medications
* Mild to moderate symptomatic asthma as defined by an Asthma Control Questionnaire score of 1.25 or greater.

Exclusion Criteria:

* Diagnosed co-morbid disease for which there are already established exercise guidelines i.e., cardiac disease or COPD
* Any other medical condition that confers greater illness morbidity than asthma (e.g., active cancer) which will confirmed by physician review
* FEV1 lower than 60% of predicted
* Incapable of exercising
* A BMI > 30 kg/m2
* Unable to speak or understand either French or English
* <18 years of age
* Patients who are currently pregnant or intend to become pregnant over the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-01; Primary Completion 2013-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Asthma control Questionnaire (Juniper) | Within 1 week of completion of the intervention (i.e., after 12 weeks)

SECONDARY OUTCOMES:
Asthma quality of life questionnaire (Juniper) | Within 1 week of completion of the intervention (i.e., after 12 weeks)
Asthma control test | Within 1 week of completion of the intervention (i.e., after 12 weeks)
Inflammatory markers | Within 1 week of completion of the intervention (i.e., after 12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Simon L Bacon, PhD, Principal Investigator — Hopital du Sacre-Coeur de Montreal / Concordia University
Locations (3):
- Canada (3):
  - Montreal Chest Institute, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec

REFERENCES:
- [Derived] Bacon SL, Lavoie KL, Bourbeau J, Ernst P, Maghni K, Gautrin D, Labrecque M, Pepin V, Pedersen BK. The effects of a multisite aerobic exercise intervention on asthma morbidity in sedentary adults with asthma: the Ex-asthma study randomised controlled trial protocol. BMJ Open. 2013 Jun 20;3(6):e003177. doi: 10.1136/bmjopen-2013-003177. PMID 23794569
- See also: PI's homepage — http://mbmc-cmcm.ca
- See also: Research Centre, Hopital de Sacre-Coeur de Montreal's homepage — http://www.crhscm.ca/